CLINICAL TRIAL: NCT03712384
Title: Personal Recovery of Young Adults With Severe Anorexia Nervosa During Adolescence: a Pilot Qualitative Study
Brief Title: Severe Anorexia Nervosa Personal Recovery
Acronym: ANAPR
Status: Completed | Type: Observational
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Other Study IDs: PSY-2014-04
Record Dates: First submitted 2018-10-15; First posted 2018-10-19 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Anorexia Nervosa; Eating Disorder
Keywords: Recovery; Qualitative research; Personal narratives
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young adult with severe anorexia: Young adult with severe Anorexia hospitalized during adolescence at Institut Mutualiste Montsouris
  Interventions: Other: Semi structured face to face interview

INTERVENTIONS:
Other: Semi structured face to face interview — Face-to-face semi-structured interview conducted in the hospital, where young adults were hospitalized 10 years before, in a quiet and isolated office. The topic guide was built according to literature review, without further change after pilot test. Interviews where audio-recorded and transcribed

SUMMARY:
A growing qualitative literature about personal recovery process in mental disorders emerges. However in Anorexia Nervosa (AN), it remains few understood, especially in severe AN during adolescence.

This pilot study seeks to enhance understanding of recovery from AN in France and support the dissemination of the PR paradigm among the French mental health community working with AN, as a complement to the medical approach.

A qualitative research according to Interpretative Phenomenological Analysis (IPA) method was conducted .Five young women hospitalized ten years before for a severe AN during their adolescence were interviewed with a semi-structured face-to-face interview on recovery process.

DETAILED DESCRIPTION:
Anorexia Nervosa (AN) is one of the most severe mental disorders with a mortality and high risk of developing chronicity. Lifetime prevalence is evaluated among women between 1.2% and 2.2%, with the higher incidence during adolescence. Recovery process remains poorly understood.

In scientific literature, recovery process of mental disorders can be seen in two different ways: the medical and the personal recovery (PR). The medical recovery is based on objective criteria, including cure (symptom disappearance), remission (symptom suspension) or therapeutic response (change of values after treatment). This medical recovery is generally studied in quantitative outcome studies. The experiential or PR is based on first person qualitative research or consensus methods, starting from patients' struggle for regaining place in their own recovery. It has become the paradigm orientation of mental health policy in anglophone countries.

A recent systematic review summeries relapse, remission or recovery criteria used in a AN outcome studies in 1-weigh measurement only; 2-symptoms reported only; 3-on both. In addition to weigh, other criteria are noticed: menstruations, psychological and behavioral features, disparities of time remission/recovery.

However, despite numerous quantitative studies, reasons for recovery, relapse or following struggle steal unclear. Medical framework is sometimes considered as reductive Moreover, those researches usually focus on risk factors, hiding protector's factors that are central for supporting recovery. Furthermore, symptom improvement is not always priority of patients(9), while improvement might happen despite symptoms persistence. Discrepancies are described in the negotiated link clinicians-patients: patient might wait for more singular and subjective approach whereas clinicians would be more invested in objective and rigorous features.

A recent systematic review offers a theorical framework to study PR in mental disorders. It is defines as an active, individual, unique, non-linearn, multidimensional and gradual process. It can be described as phase or stage, as struggle, as a life-changing experience or even as a trial or error process. It may be structured by a turning point, after when there are no turning back. It is aided by supporting and healing environment, and might occur without cure. Starting from first person narratives of mental disorders recovery, five factors supporting recovery are described: connectedness, hope and optimism about the future, identity, meaning in life, empowerment. One meta-ethnography review was published on qualitative research about PR in AN, concerning 8 studies. It provides elements on process of change, factors supporting PR and notion of empowerment and self-reconciliation.

Finally, most of PR studies come from USA, UK, Australia and Canada. Further research are needed to ground PR including cultural context. In France, AN PR has been rarely studied. These study tries to enhance understanding AN recovery in French context, to support implementation of PR paradigm among French mental health AN community; complementary to medical approach.

Study questions are: how people who suffered of severe AN and experienced hospitalization during adolescence feel and make sense to their recovery?

METHODS This study is a qualitative research with IPA, supplemented by quotation of ICD 10 criteria. We reported COREQ 32 guidelines.

Setting and participants IPA recommends homogeneous and short sampling so as to better appreciate convergences and divergences of phenomena. To maximize homogenization, very precise criteria (presented in box 1) were first chosen in order to focus on studied phenomena with in-depth way, before opening to wider study on AN recovery. Recruitment was restrained to the same hospital (Institut Mutualiste Montsouris) at the same year of hospitalization, so as to homogenize experience of care. Period of 10 years was chosen for being widely beyond largest literature mean criteria of medical recovery fixed at seven years, to get some distance with recovery process.

ELIGIBILITY:
Inclusion Criteria:

* woman
* Adult between 20 and 30 years old
* With history of restrictive AN (CIM 10: F50)
* Without no other comorbidity
* Hospitalized for AN during adolescence (10-19 years old) ten years ago, in adolescent psychiatry at Institute Mutualiste Montsouris (France)
* Native French speaker
* Considers herself recovered
* Agreement

Exclusion Criteria:

* Presence of AN criteria (ICD-10: F50) during research interview,
* Absence of all recovery qualitative criteria after qualitative analysis

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young people who suffered of severe AN and experienced hospitalization during adolescence feels recovered
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-06-20 (Actual); Primary Completion 2014-07-05 (Actual); Study Completion 2014-07-05 (Actual)

PRIMARY OUTCOMES:
Recovery process of AN | Semi structured face to face interview, 10 years after hospitalization for AN.
  Initial interview topic guide domain
  1. How have you spent your life for the first hospitalization for AN?
  2. What are the factors that help or prevent from going ahead?
  3. All this way long, how did feel talking about yourself?
  4. How did evolve your relationships?
  5. How have you felt your body all this way long?
  6. How do you define recovery of AN during adolescence?
  7. How would you define yourself?
  8. What kind of stories do you tell yourself about AN?
  9. If you would be faced with someone with current AN, what would you advice him/her?

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Aude PIOT, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Institut mutualiste montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khalsa SS, Portnoff LC, McCurdy-McKinnon D, Feusner JD. What happens after treatment? A systematic review of relapse, remission, and recovery in anorexia nervosa. J Eat Disord. 2017 Jun 14;5:20. doi: 10.1186/s40337-017-0145-3. eCollection 2017. PMID 28630708
- [Background] Arcelus J, Mitchell AJ, Wales J, Nielsen S. Mortality rates in patients with anorexia nervosa and other eating disorders. A meta-analysis of 36 studies. Arch Gen Psychiatry. 2011 Jul;68(7):724-31. doi: 10.1001/archgenpsychiatry.2011.74. PMID 21727255
- [Background] Strober M, Freeman R, Morrell W. The long-term course of severe anorexia nervosa in adolescents: survival analysis of recovery, relapse, and outcome predictors over 10-15 years in a prospective study. Int J Eat Disord. 1997 Dec;22(4):339-60. doi: 10.1002/(sici)1098-108x(199712)22:43.0.co;2-n. PMID 9356884
- [Background] Leamy M, Bird V, Le Boutillier C, Williams J, Slade M. Conceptual framework for personal recovery in mental health: systematic review and narrative synthesis. Br J Psychiatry. 2011 Dec;199(6):445-52. doi: 10.1192/bjp.bp.110.083733. PMID 22130746
- [Background] Wollburg E, Meyer B, Osen B, Lowe B. Psychological change mechanisms in anorexia nervosa treatments: how much do we know? J Clin Psychol. 2013 Jul;69(7):762-73. doi: 10.1002/jclp.21945. Epub 2013 Jan 24. PMID 23349069
- [Background] Espindola CR, Blay SL. Anorexia nervosa's meaning to patients: a qualitative synthesis. Psychopathology. 2009;42(2):69-80. doi: 10.1159/000203339. Epub 2009 Feb 19. PMID 19225241
- [Background] Noordenbos G, Seubring A. Criteria for recovery from eating disorders according to patients and therapists. Eat Disord. 2006 Jan-Feb;14(1):41-54. doi: 10.1080/10640260500296756. PMID 16757448
- [Background] Westwood LM, Kendal SE. Adolescent client views towards the treatment of anorexia nervosa: a review of the literature. J Psychiatr Ment Health Nurs. 2012 Aug;19(6):500-8. doi: 10.1111/j.1365-2850.2011.01819.x. Epub 2011 Sep 27. PMID 22070426
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Jenkins J, Ogden J. Becoming 'whole' again: a qualitative study of women's views of recovering from anorexia nervosa. Eur Eat Disord Rev. 2012 Jan;20(1):e23-31. doi: 10.1002/erv.1085. Epub 2011 Mar 10. PMID 21394835